CLINICAL TRIAL: NCT06406946
Title: Investigating the Effects of Lions Mane Mushroom, and a Mushroom Blend on Wellbeing in Stressed/Anxious Gen Z Women
Brief Title: Mushrooms, Mood and Mental Wellbeing in Gen Z Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65CG2
Record Dates: First submitted 2024-04-17; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Well-Being, Psychological; Mood; Anxiety; Stress
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lions Mane (Experimental): Lion's mane (1.8 gram per day, consisting of 3 x 600mgcapsules)
  Interventions: Dietary Supplement: Lion's mane blend
- Mushroom Blend (Experimental): Lion's mane and reishi mushroom blend (1.8 gram per day, consisting of 3x600mg capsules)
  Interventions: Dietary Supplement: Lion's mane and reishi blend
- Placebo (Placebo Comparator): (1.8-gram microcrystalline cellulose placebo powder, 3x600mg capsules).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lion's mane blend — 1.8 gram per day of lions mane, consisting of 3 x 600mg capsules
  Arms: Lions Mane
Dietary Supplement: Lion's mane and reishi blend — 1.8 gram per day of lions mane and reishi blend, consisting of 3 x 600mg capsules
  Arms: Mushroom Blend
Dietary Supplement: Placebo — 1.8-gram microcrystalline cellulose placebo powder, 3x600mg capsules
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effects of 28 days supplementation of Lions mane mushroom and mushroom blend of Lions mane and reishi mushroom, on wellbeing in stressed or anxious women.

The study will follow a randomized, double-blind, placebo-controlled, parallel group design. Participants will receive either lion's mane mushroom mane (1.8 gram per day, consisting of 3 x 600mgcapsules), a blend of lion's mane mushroom and reishi mushroom 1.8 gram per day, consisting of 3x600mg capsules) or placebo (1.8-gram microcrystalline cellulose placebo powder, 3x600mg capsules).

The trial will utilise Generalised Anxiety Disorder Assessment (GAD-7); the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS); Chalder Fatigue Scale; Rosenberg's Self-Esteem Scale; Perceived Stress Scale (PSS) and Stress Visual Analogue Scales (S-VAS) at baseline and after 28 days supplementation. Participants will complete the HADS and S-VAS at home on days 7, 14 and 21. On day 42 (14 days after treatment ending) participants will complete the GAD-7, HADS and S-VAS.

135 healthy women (who self-report being stressed and/or anxious) aged 18-26 (and born between 1997 and 2013) will be recruited using opportunity sampling. Participants will be supplied with either one of the active treatments or the placebo (allocated by a randomised schedule) whilst visiting the research centre for the testing appointments and will take treatment home to consume daily for the duration of the study. Participants will record time of taking treatment each day in a treatment diary which will be returned to the research centre, along with any unused treatment, upon completion of the study.

DETAILED DESCRIPTION:
The study will follow a randomized, double-blind, placebo-controlled, parallel group design. Participants will receive either lion's mane, a blend of lion's mane mushroom and reishi mushroom or placebo to be consumed at home each day.

Participants will initially attend a virtual screening session (conducted via telephone call or Microsoft Teams), this session will involve:obtaining of informed consent, health screening, completion of the Caffeine Consumption Questionnaire (CCQ) and collection of demographic information. Participants will then attend testing labs on two occasions.

The first session will take place at an agreed time, with no restrictions to the participant in terms of abstinence from caffeine, food etc - participants will be encouraged to follow their normal routine and to also do this prior to completing the other assessments. This session will comprise collection of physiological measures that cannot be completed remotely (blood pressure, height and weight,waist-hip-ratio). Participants will then complete the baseline wellbeing questionnaires: Generalised Anxiety Disorder Assessment (GAD-7); the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS); Chalder Fatigue Scale; Rosenberg's Self-Esteem Scale; Perceived Stress Scale (PSS) and Stress Visual Analogue Scales (S-VAS). Participants will receive their treatment, they will be instructed to consume 3 capsules per day for the next 28-days. This appointment will take ~30 mins.

At home on Days 7, 14 and 21 participants will complete interim mood questionnaires. During these they will complete the HADS and S-VAS only.

On Day 28, participants will return to the laboratory to complete their final wellbeing assessment in person. This is the full wellbeing assessment as completed on Day 1. During this visit participants will also return their unused treatment and complete a treatment guess form. Participants will also provide qualitative (written) feedback on if they felt any changes in their mood/wellbeing during the course of the trial.

To assess if there are any wellbeing changes following ceasing consumption of treatment, participants will also complete a final wellbeing assessment on Day 42 (14 days after treatment ending). For this assessment they will complete the GAD-7, HADS and SVAS, alongside the qualitative feedback on any observed changes since stopping the treatment.

A sample of 135 women aged 18-26 (born between 1997-2013) who feel that they are anxious and/or stressed (but with no diagnosis of a psychiatric disorder) will be recruited from the North East area to take part in this study. Participants will be randomly allocated to one of the active treatments, or placebo, neither the participant nor the researcher will know which group they have been allocated to.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a woman
* Are aged 18 to 26 years at the time of giving consent (to be classified as Gen Z participants must have been born 1997-2013)
* Rate themselves as stressed and/or anxious
* Be a native speaker of English or fluent in English

Exclusion Criteria:

* Have any pre-existing medical condition/illness which will impact taking part in the study. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance NOTE: the explicit exceptions to this is controlled hayfever, asthma, hypo/hyperthyroidism, high blood pressure, high cholesterol, reflux, dyslexia/dyscalculia, ADHD, autism.
* Are currently taking prescription medications (NOTE: the explicit exceptions to this are contraceptive treatments for female participants, and those taken 'as needed' in the treatment of asthma and hay fever. There may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening). Within this trial medication for diagnosed neurological conditions (e.g. ADHD) will be allowed as long as medication has been taken for a minimum of 3 months and will be taken consistently throughout the trial period.
* Have relevant food allergies/ intolerances/ sensitivities
* Excessive caffeine intake (> 500 mg per day)
* Have taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taken are out of choice and not medically prescribed or advised. NOTE - Vitamin D and iron supplements are allowed for this trial if they have been advised by GP to increase levels to a normal range and have been taken for at least 4 weeks consistently and will be taken consistently throughout the trial.
* Are pregnant, seeking to become pregnant or lactating
* Have taken antibiotics within the past 4 weeks
* Are currently participating in other clinical or nutrition intervention studies, or have done so in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months (this includes medically diagnosed anxiety and depression)
* Suffer from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Have any known active infections
* Will be non-compliant with treatment consumption

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must identify as a woman
Enrollment: 135 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline, following 28 days supplementation and 14 days after ceasing supplementation
  Ratings of anxiety measured via the Generalised Anxiety Disorder Assessment (GAD-7). The outcome of the questionnaire is reported as a score between 0 and 21, with 0 indicating no anxiety and 21 indicating the highest level of anxiety. Scores are clinically categorised as: 0-4 (none), 5-9 (mild), 10-14 (moderate) and 15-21 (severe).

SECONDARY OUTCOMES:
Anxiety | Baseline, following, 7, 14, 21 and 28 days supplementation and 14 days after ceasing supplementation
  Ratings of anxiety measured via the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS). The outcome of the anxiety subscale is reported as a score between 0 and 21. With scores divided into four stages: 0-7 (Normal), 8-10 (Mild), 11-15 (Moderate), 16-21 (Severe).
Stress | Baseline and following 28 days supplementation
  Ratings of stress measured via the Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40, with higher scores indicating higher perceived stress. Scores 0-13 are considered low stress; 14-26 considered moderate stress; 27-40 considered high stress.
Stress | Baseline, following, 7, 14, 21 and 28 days supplementation and 14 days after ceasing supplementation
  Subjective feelings of stress using Stress Visual Analogue Scales. Participants complete 4 visual analogue scales assessing how anxious, stressed, relaxed and calm they feel (Not at all (0) - Extremely (100)). An average 'stress' score is created using this data, this score ranges from 0 to 100, with a higher score indicating higher perceived stress.
Fatigue | Baseline and following 28 days supplementation
  Subjective feelings of fatigue using the Chalder Fatigue Scale. Using Likert style scoring, individuals score in a range from 0 to 33. With a higher score indicating higher levels of fatigue.
Self Esteem | Baseline and following 28 days supplementation
  Ratings of self esteem using Rosenbergs Self Esteem Scale. An individual will score from 0 to 30. With a lower score indicating lower self esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Docherty, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided